CLINICAL TRIAL: NCT03531775
Title: Upright Magnetic Resonance Imaging in COPD and Diaphragm Disease
Brief Title: Upright MRI in Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Shahideh Safavi, Principal Investigator, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18011
Record Dates: First submitted 2018-04-27; First posted 2018-05-22 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: COPD With Hyperinflation; Diaphragmatic Weakness
Keywords: upright MRI; COPD with hyperinflation; Diaphragmatic weakness

STUDY DESIGN:
Intervention Model Description: Clinical trial to study a novel intervention (upright MRI) to compare interventions in clinical practice
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upright MRI (Other): All participants will be scanned using an upright MRI in seated/standing position and supine position. They will also be scanned supine using a conventional MRI.
  Interventions: Diagnostic Test: Upright MRI

INTERVENTIONS:
Diagnostic Test: Upright MRI — Participants will be scanned using an upright MRI in sitting/standing position and supine position. They will also be scanned in supine position using a conventional MRI.

SUMMARY:
The diaphragm is the main muscle assisting breathing. This study aims to assess the use of MRI in patients with diaphragmatic weakness and patients with Chronic Obstructive Pulmonary Disease (COPD) who have hyperinflation. In some patients with COPD, air gets trapped in the lungs and causes them to expand too much; this is called hyperinflation. These patient report severe breathlessness, which may be in part because of their diaphragm. It is known that posture impacts lung function and breathing and the investigators want to assess the effect of posture on the diaphragm. Currently, lung function tests and CT or ultrasound scan are the main tests used to check how the diaphragm works. Recently, at University of Nottingham, an new imaging approach has been developed that uses an upright MRI allowing testing the patients in lying position and seated/standing in the same scanner. This may help researchers test the diaphragm position and shape more accurately and check the effects of posture on the diaphragm. This may help researchers and clinicians better understand the relationship between postural changes in diaphragm position and shape and symptoms.

The study will take place at the clinical research MRI centre at Nottingham Medical School, which is next to Queen's Medical Centre. The investigators want to recruit healthy volunteers, patients with diaphragmatic weakness and patients with COPD whose lungs are hyperinflated. The study will last 2 years, and the participants are asked to attend the imaging centre only once, where they will give consent and will be scanned at the same visit, which is expected to take 2 hours to complete. They will be scanned on two scanners: lying and seated/standing in the new upright scanner and lying in a conventional scanner. The investigators will not use any contrast for imaging, i.e. participants will not be injected with a dye and they will breathe air.

DETAILED DESCRIPTION:
This is a single centre, proof of concept clinical trial. The investigators want to recruit healthy volunteers, patients with diaphragmatic weakness and patients with COPD whose lungs are hyperinflated. Half the investigators are clinicians and have asked their patient whether such a study would interest them, and patients have been very supportive. This study addresses an unanswered clinical question.

The participants will be adults, men and women, who can give informed consent, and can cooperate with the study procedures. As the participants will be scanned using MRI, people who are unsuitable for MRI scanning, for example those with a pacemaker, will be excluded from the study for safety reasons.The participant will be observed by a clinical investigator throughout the study visit.

As for side effects / risks, no medicinal products will be administered in this study. Some participants may experience anxiety while undergoing MRI scan. It is expected that some patients may not be able to lie flat in the scanner, in which case they will be asked only to undergo scans that they are able to tolerate.

In addition to being scanned using an upright MRI and a conventional MRI, the following measurements will be takes: weight, height, blood pressure, heart rate, oxygen saturation, respiratory rate, and spirometry. The participants will be asked to fill a St George's Respiratory Questionnaire and an MRC (Medical Research Council) Dyspnoea Scale. A detailed medical history will be taken.

The participants will be assigned unique codes, and their data will be anonymised. Participants' medical reports will only be accessed for study purposes and will be treated as confidential.

The investigators will aim to use the data to plan future studies, and the data from this study may contribute to publications and presentations. Participants will not be identified in any publications arising from the research. The data obtained will be published without any identifying information..

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  * Adult - Male or female, aged 18 to 90 years old
  * Capacity to give informed consent
  * Able to hold their breath for 10 seconds
  * Able to understand the requirements of the study and to cooperate with the study procedures
* Cohort-specific inclusion criteria:

Healthy participants

* No reported or diagnosed chronic respiratory disease

COPD with hyperinflation

* Evidence of airflow obstruction on spirometry - FEV1/FVC < 0.7 and FEV1 <80%. (FEV1 = full expiratory volume in 1 second, FVC = full vital capacity)
* Diagnosis of hyperinflation based on imaging or lung function measures.

Diaphragm weakness due to non-neuromuscular disease

* Established diagnosis of diaphragm weakness due to non-neuromuscular disease, e.g. viral illness, trauma.

Diaphragm weakness due to neuromuscular disease

* Established diagnosis of diaphragm weakness due to neuromuscular disease

Exclusion Criteria:

* Unsuitable for MRI scanning (e.g. have metal implants/pacemaker or contraindicated following questionnaire)
* Deemed unlikely to comply with instructions during imaging
* Deemed not fit enough to tolerate procedure
* Deemed unsuitable by clinical investigator for other reasons
* History of lung volume reduction procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-16 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The diaphragm will be imaged using MRI in horizontal and vertical positions. | 2 years
  Images will be anonymised and stored securely on University servers.
The change in diaphragm position and morphology on MRI following a change in posture (vertical to horizontal position or vice versa) will be measured. | 2 years
The diaphragm position and morphology in COPD patients with hyperinflation will be imaged using MRI. | 2 years
The diaphragm position and morphology in patients known to have diaphragmatic weakness will be imaged using MRI. | 2 years

SECONDARY OUTCOMES:
The lung function abnormality will be compared with abnormalities in diaphragm position and morphology as noted on MRI. | 2 years
The patients' symptoms, as reported on St George's Respiratory Questionnaire and a visual analogue scale for breathlessness, will be compared to the abnormalities noted in diaphragm position and morphology on MRI. | 2 years
  Participants will be asked to fill St George's Respiratory questionnaire and a visual analogue scale for breathlessness to assess symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shahideh Safavi, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham
  - University of Nottingham, Nottingham